CLINICAL TRIAL: NCT00505414
Title: A Randomized Withdrawal, Active- and Placebo-controlled, Double-blind, Multi-center Phase III Trial Assessing Safety and Efficacy of Oral CG5503 (Tapentadol) Prolonged Release (PR*) in Subjects With Moderate to Severe Chronic Malignant Tumor-related Pain. *Prolonged Release and is the Recommended Nomenclature for Use in the European Union (EU). ER Means Extended Release and is the Recommended Nomenclature for Use in the United States of America (USA). "PR" is Synonymous With "ER" and is Interchangeable.
Brief Title: A Study to Evaluate the Effectiveness and Safety of CG5503 (Tapentadol) in the Treatment of Chronic Tumor Related Pain Compared With Placebo and Morphine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recall of rescue medication, alternative rescue medication availability issues.
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 672519; 2007-001985-34 (EudraCT Number); KF5503/16 (Other: Grünenthal GmbH)
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pain; Neoplasm; Cancer
Keywords: Chronic Tumor Related Pain; Analgesic; Tapentadol Extended Release; Morphine Sulfate Controlled Release; Pain assessment; Placebo
MeSH Terms: conditions — Pain; Neoplasms | interventions — Tapentadol; Morphine; Masks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matching Placebo (Placebo Comparator): Oral Tapentadol 100 mg to 250 mg twice daily. Followed by matching placebo in the maintenance (i.e. randomized withdrawal phase).
  Interventions: Drug: Matching Placebo in the Maintenance Phase after Tapentadol in the Titration Phase
- Morphine Controlled Release (Active Comparator): Oral Morphine 45 mg to 90 mg twice daily.
  Interventions: Drug: Morphine in the Maintenance Phase; Drug: Morphine in the Titration Phase
- Tapentadol Extended Release (Experimental): Oral Tapentadol 100 mg to 250 mg twice daily.
  Interventions: Drug: Tapentadol in the Titration Phase; Drug: Tapentadol in the Maintenance Phase

INTERVENTIONS:
Drug: Tapentadol in the Titration Phase
  Other Names: Palexia; Nucynta
  Arms: Tapentadol Extended Release
Drug: Morphine in the Maintenance Phase — Participant started the trials with 45 mg morphine controlled release twice daily. Upward titration could then occur at a minimum of 3-day intervals in increments of 15 mg morphine twice daily. The maximum dose of morphine controlled release was 90 mg twice daily. Downward titration (but not below 45 mg twice daily) was permitted. In the maintenance phase participants continued on the dose level established in titration phase.
  Participants randomized to the morphine arm remained on morphine if they qualified for the maintenance phase of the study. The participants were maintained on the dose established at the end of the titration phase. The adverse events listed were documented in the maintenance phase.
  Other Names: MS Contin overencapsulated for blinding
  Arms: Morphine Controlled Release
Drug: Matching Placebo in the Maintenance Phase after Tapentadol in the Titration Phase — Participant randomized to placebo in the maintenance phase received 100 mg tapentadol prolonged release twice daily for 3 days to taper them off of the tapentadol dose they had received in the titration period. From the fourth day of the maintenance period onwards they received placebo twice daily.
  Arms: Matching Placebo
Drug: Tapentadol in the Maintenance Phase — The participants re-randomized to receive tapentadol prolonged release in the maintenance phase were maintained on the dose established in the titration phase.
  Arms: Tapentadol Extended Release
Drug: Morphine in the Titration Phase — After signing informed consent eligible subjects were randomized to receive morphine controlled release. The oral medication was taken twice daily, morning and evening every 12 hours (with a minimum of 6 hours between doses). Participant started the trials with 45 mg morphine controlled release twice daily. Upward titration could then occur at a minimum of 3-day intervals in increments of 15 mg morphine twice daily. The maximum dose of morphine controlled release was 90 mg twice daily. Downward titration (but not below 45 mg twice daily) was permitted.
  Arms: Morphine Controlled Release

SUMMARY:
The purpose of this study is to determine whether CG5503 (tapentadol) is effective and safe in the treatment of chronic tumor related pain compared to placebo.

DETAILED DESCRIPTION:
Normally chronic tumor related pain is controlled when subjects receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. Tapentadol, a newly synthesized drug with an Prolonged Release (ER) formulation, also acts as a centrally acting pain reliever but has a dual mode of action.

The aim of this trial is to investigate the effectiveness (level of pain control) and safety (side effects) of Tapentadol Prolonged Release (ER) compared to a tablet with no active ingredient drug (placebo) and a corresponding dose of Morphine (an opioid commonly used to treat tumor related pain). This trial is a randomized, double-blind (neither investigator nor patient will know which treatment was received), active- and placebo-controlled, parallel-group, randomized-withdrawal, multicenter trial. To maintain the blind all subjects were re-randomized at the start of the maintenance period. To maintain the blind all tapentadol subjects were re-randomized at the start of the maintenance period. Subjects that received morphine in the titration period continued in the maintenance period on morphine.

The trial includes a 2 week titration phase starting with either 45 mg Morphine Sulfate Controlled Release (CR) twice daily or 100 mg tapentadol ER taken twice daily (bid). Based on effectiveness and side effects participants can up-titrate in steps of 50 mg Tapentadol ER or 15 mg Morphine Sulfate CR to a maximal dose of 250 mg Tapentadol ER bid or 90 mg Morphine Sulfate CR twice daily respectively. If subjects meet the stabilization criteria at the end of the titration phase they will be re-randomized to either placebo or active treatment and will continue 4 weeks at the last dose level in the maintenance phase.

Assessments of pain relief, defined as a responder include the pain intensity numeric rating scale (NRS). The Patient Global Impression of Change scale (PGIC) will also be used as a secondary efficacy endpoint. Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of tapentadol.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent document.
* Male and non-pregnant, non-lactating female subjects.
* Female subjects must be post menopausal, surgically sterile, or practicing an effective method of birth control and continue to do so throughout the trial.
* At least 18 years of age.
* Have chronic malignant tumor-related pain
* Are opioid-naïve or have been pretreated with an equianalgesic dose range equivalent of up to 160 mg oral morphine per day and are dissatisfied with prior treatment.
* Have a mean pain intensity of at least 5 points on an 11-point Numeric Rating Scale (where 0 indicates no pain and 10 indicates worst possible pain).
* Have an expected course of the disease such that the pain that will permit compliance with the trial protocol over the entire trial period.

Exclusion Criteria:

* Have a life-long history of seizure disorder or epilepsy.
* Have had any of the following within one year: mild/moderate traumatic brain injury, stroke, and transient ischemic attack.
* Have had severe traumatic brain injury within 15 years (consisting of ≥ 1 of the following: brain contusion, intracranial hematoma, and either unconsciousness or post-traumatic amnesia lasting for more than 24 hours) or residual sequelae suggesting transient changes in consciousness.
* Have a known history and/or presence of cerebral metastases.
* Have moderately or severely impaired hepatic function.
* Have laboratory values reflecting inadequate hepatic function.
* Have thrombopenia, leucopenia or hypercalcemia
* Have severely impaired renal function.
* Having uncontrolled hypertension
* Having clinically relevant history of hypersensitivity, allergy or contraindications to morphine or any of the excipients.
* Have chronic hepatitis B or hepatitis C, or Human Immunodeficiency Virus (HIV).
* Subjects currently undergoing the following concomitant therapy: radiotherapy, pain inducing chemotherapy, anti-parkinsonian drugs, neuroleptics, monoamine oxidase inhibitors, serotonin norepinephrine re-uptake inhibitors (SNRI) or any other analgesic therapy than investigational medication or rescue medication during the trial. Selective serotonin re-uptake inhibitor (SSRI) treatments are allowed if taken for at least 30 days before the screening period of the trial at an unchanged dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Poulain, Dr., Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (37):
- United States (7):
  - 001013, St. Petersburg, Florida
  - 001002, Elkhart, Indiana
  - 001001, Shreveport, Louisiana
  - 001010, Cedarhurst, New York
  - 001003, Glens Falls, New York
  - 001004, Winston-Salem, North Carolina
  - 001015, Canton, Ohio
- Argentina (9):
  - 054003, La Plata, Buenos Aires
  - 054012, Pergamino, Buenos Aires
  - 054022, Quilmes, Buenos Aires
  - 054008, Villa Domínico, Buenos Aires
  - 054010, Rosario, Santa Fe Province
  - 054013, Rosario, Santa Fe Province
  - 054005, San Miguel de Tucumán, Tucumán Province
  - 54009, Ciudad de Buenos Aires
  - 054015, Santa Fe
- Chile (7):
  - 056006, Coquimbo
  - 056011, Santiago
  - 056008, Santiago
  - 056005, Santiago
  - 056003, Talcahuano
  - 056004, Temuco
  - 056012, Valparaíso
- France (3):
  - 033002, Nice
  - 033015, Orléans
  - 033001, Villejuif
- Latvia (2):
  - 371001, Daugavpils
  - 371002, Riga
- Ukraine (9):
  - 380015, Cherkasy
  - 380011, Donetsk
  - 380012, Donetsk
  - 380008, Kharkiv
  - 380002, Kharkiv
  - 380013, Kiev
  - 380001, Kiev
  - 380009, Lviv
  - 380010, Poltava

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant in was enrolled on 29 June 2007 and the Last participant out was on the 02 February 2009. In general this was an out-patient study subject to country specific regulations.
Pre-assignment Details: Eligible participants were required to stop their previous analgesic [pain treatment] therapy at randomization. 136 participants consented. 43 participants were not eligible for randomization to tapentadol extended release or morphine controlled release at baseline. 93 participants started the titration period.
Groups:
- Morphine (Maintenance Phase): Participants in the maintenance phase continued on the dose level established in titration phase, i.e. 45 mg to 90 mg twice daily.
- Tapentadol (Maintenance Phase): Participants re-randomized to tapentadol prolonged release in the maintenance phase continued on the dose level established at the end of the titration phase. Oral tapentadol 100 mg to 250 mg twice daily.
- Matching Placebo (Maintenance Phase): Participants were re-randomized to placebo after being on tapentadol in the titration phase. At the start of this phase participants received 100 mg tapentadol prolonged release twice daily for 3 days to taper them off of the tapentadol dose they had received in the titration period. From the fourth day of the maintenance period onwards they received placebo twice daily.
- Tapentadol (Titration Phase): After signing informed consent eligible participants were randomized to receive tapentadol extended release. Oral tapentadol 100 mg up to 250 mg twice daily. The oral medication was taken twice daily, morning and evening every 12 hours (with a minimum of 6 hours between doses).
- Morphine (Titration Phase): After signing informed consent eligible participants were randomized to receive morphine controlled release. The oral medication was taken twice daily starting at 45 mg up to 90 mg twice daily, morning and evening every 12 hours (with a minimum of 6 hours between doses).
Period: Titration Phase
Arm/Group | Morphine (Maintenance Phase) | Tapentadol (Maintenance Phase) | Matching Placebo (Maintenance Phase) | Tapentadol (Titration Phase) | Morphine (Titration Phase)
Started | 0 | 0 | 0 | 62 | 31
Completed | 0 | 0 | 0 | 32 | 19
Not Completed | 0 | 0 | 0 | 30 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 8 | 3
Not completed — Death | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 10 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 4
Not completed — Underlying disease and therapy required | 0 | 0 | 0 | 7 | 3
Period: Maintenance Phase
Arm/Group | Morphine (Maintenance Phase) | Tapentadol (Maintenance Phase) | Matching Placebo (Maintenance Phase) | Tapentadol (Titration Phase) | Morphine (Titration Phase)
Started | 18 (18 of the 19 morphine participants continued with morphine in the maintenance phase.) | 15 (15 of 32 tapentadol titration participants continued with tapentadol in the maintenance phase) | 14 (14 of 32 tapentadol titration participants were treated with placebo in the maintenance phase.) | 0 (29 of 32 participants were treated in the maintenance phase either with placebo or tapentadol) | 0 (18 of 19 participants completing the morphine titration phase were continued on morphine.)
Did Not Qualify for Maintenance Phase | 0 | 0 | 0 | 3 | 1
Completed | 12 | 10 | 6 | 0 | 0
Not Completed | 6 | 5 | 8 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 3 | 0 | 0
Not completed — Death | 2 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — underlying disease and therapy required | 0 | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set. The information is correct for each treatment arm. The demographic details for the total population is for the 93 participants that started treatment in the titration phase of the trial.
  The tapentadol titration population was subject to a randomized withdrawal-trial design in the maintenance phase.
Groups:
- Tapentadol (Titration Phase): After signing informed consent eligible participants were randomized to receive tapentadol extended release. Oral tapentadol 100 mg to 250 mg twice daily. The oral medication was taken twice daily, morning and evening every 12 hours (with a minimum of 6 hours between doses).
- Morphine (Titration Phase): After signing informed consent eligible subjects were randomized to receive morphine controlled release. The oral medication was taken twice daily starting at 45 mg up to 90 mg twice daily, morning and evening every 12 hours (with a minimum of 6 hours between doses).
- Total: Total of all reporting groups
Arm/Group | Tapentadol (Titration Phase) | Morphine (Titration Phase) | Total
Number analyzed (Participants) | 62 | 31 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Not all participants of the titration phase participated in the maintenance phase. The tapentadol titration population was subject to a randomized withdrawal-trial design in the maintenance phase and received either tapentadol or placebo.
  years
    Titration Phase | 62.4 (12.51) | 60.6 (11.77) | 61.8 (12.23)
    Tapentadol Maintenance: number analyzed (Participants) | 15 | 0 | 15
    Tapentadol Maintenance | 63.5 (9.34) |  | 63.5 (9.34)
    Placebo Maintenance: number analyzed (Participants) | 14 | 0 | 14
    Placebo Maintenance | 61.0 (12.93) |  | 61.0 (12.93)
    Morphine Maintenance: number analyzed (Participants) | 0 | 18 | 18
    Morphine Maintenance |  | 58.4 (12.65) | 58.4 (12.65)
Sex/Gender, Customized [Number; unit: participants]
  Female (Titration) | 35 | 12 | 47
  Male (Titration) | 27 | 19 | 46
  Female (Morphine (Maintenance) | 0 | 8 | 8
  Male (Morphine Maintenance) | 0 | 10 | 10
  Female (Tapentadol Maintenance) | 9 | 0 | 9
  Male (Tapentadol Maintenance) | 6 | 0 | 6
  Female (Placebo Maintenance) | 8 | 0 | 8
  Male (Placebo Maintenance) | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 41 | 19 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 11 | 32
Region of Enrollment [Number; unit: participants]
  France | 5 | 0 | 5
  United States | 3 | 4 | 7
  Argentina | 14 | 7 | 21
  Ukraine | 16 | 5 | 21
  Chile | 18 | 9 | 27
  Latvia | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Responder Rates in Maintenance Period
Description: A "responder" is a participant in the study that:
  1. completed 28 days of the maintenance phase
  2. had a numeric rating scale score below 5 on the 11 point scale (where 0 indicates no pain and 10 indicates worst possible pain. This twice daily current pain score was averaged over Day 18 to Day 43.
  3. did not use more than 30 mg of rescue medication per day on average in the 28 day (excluding the first 3 days) maintenance period (from Day 18 to Day 43).
  A participant that met all 3 of the above-mentioned criteria is counted as a responder, in other words the participant benefited from the assigned drug treatment. A participant that fails to meet at least 1 of the 3 criteria is not counted as a responder.
Time Frame: End of the 4 week Maintenance Phase (Day 43)
Population: Full Analysis Set. Number of participants with data available.
Measure: Number; unit: participants
Arm/Group | Morphine (Maintenance Phase) | Tapentadol (Maintenance Phase) | Matching Placebo (Maintenance Phase)
Number analyzed (Participants) | 18 | 15 | 14
participants | 6 | 8 | 3

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change (PGIC) is an instrument where the participant indicates their perceived change at the end of a treatment phase. The overall participant status assessed using Patient Global Impression of Change (PGIC) self-assessment questionnaire which was used by participants to report on 7 categories listed as follows; Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse and Very Much Worse in tapentadol and morphine at Day 15 (Start of Maintenance Phase) and repeated in participants completing the Maintenance Phase in the Matching Placebo, Tapentadol and Morphine (Day 43).
Time Frame: Day 15 corresponds with PGIC at end of titration phase; Day 43 corresponds with PGIC at end of maintenance phase
Population: Full Analysis Set. Number of participants with data available.
Measure: Number; unit: participants
Arm/Group | Morphine (Maintenance Phase) | Tapentadol (Maintenance Phase) | Matching Placebo (Maintenance Phase) | Tapentadol (Titration Phase) | Morphine (Titration Phase)
Number analyzed (Participants) | 18 | 15 | 14 | 62 | 31
participants
  Very Much Improved | 1 | 0 | 0 | 0 | 0
  Much Improved | 3 | 8 | 2 | 5 | 1
  Minimally Improved | 4 | 4 | 4 | 8 | 4
  No Change | 4 | 1 | 1 | 3 | 2
  Minimally Worse | 0 | 1 | 0 | 4 | 0
  Much Worse | 1 | 1 | 2 | 2 | 0
  Very Much Worse | 0 | 0 | 0 | 0 | 0
  Missing | 5 | 0 | 5 | 40 | 24

ADVERSE EVENTS:
Time Frame: Participants were to be treated for up to 42 days: Titration (14 days) and Maintenance Phase (up to 28 days).
Description: More than one event might have occured in the same participant.
Arm/Group | Morphine (Maintenance Phase) | Tapentadol (Maintenance Phase) | Matching Placebo (Maintenance Phase) | Tapentadol (Titration Phase) | Morphine (Titration Phase)
Serious Adverse Events (participants affected / at risk) | 4/18 | 2/15 | 4/14 | 11/62 | 4/31
Other Adverse Events (participants affected / at risk) | 12/18 | 9/15 | 7/14 | 28/62 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (Maintenance Phase) (N=18) | Tapentadol (Maintenance Phase) (N=15) | Matching Placebo (Maintenance Phase) (N=14) | Tapentadol (Titration Phase) (N=62) | Morphine (Titration Phase) (N=31)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 — The participant was initially in the tapentadol titration phase with the first episode of anemia. The participant was subsequently in the placebo maintenance treatment group. Participant was withdrawn. Outcome of the third event was fatal.
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 3 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental Status Change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (Maintenance Phase) (N=18) | Tapentadol (Maintenance Phase) (N=15) | Matching Placebo (Maintenance Phase) (N=14) | Tapentadol (Titration Phase) (N=62) | Morphine (Titration Phase) (N=31)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 1
Choluria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 6 | 3
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 4 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 5 | 0
Lip Oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 7 | 4
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 1 | 3 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 9 | 2

LIMITATIONS AND CAVEATS:
Early termination, due to a recall of the morphine rescue medication and issues regarding supply of an alternative, lead to only 93 participants out of the 573 planned (16%) being available for analysis. The data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor and the Sponsor's designee reserves the right to review any publication pertaining to the trial at least 30 days before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.